CLINICAL TRIAL: NCT03193411
Title: Visumax Femtolasik Versus Moria M2 Microkeratome in Mild to Moderate Myopia: Efficacy, Safety, Predictability, Aberrometric Changes and Flap Thickness Predictability
Brief Title: Visumax Femtolasik Versus Moria M2 Microkeratome in Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dar Al Shifa Hospital (Other)
Responsible Party: Principal Investigator, magda torky, priniciple investigator, Dar Al Shifa Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2315
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Lasik in Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microkeratome group (Other): 30 eyes were treated by microkeratome
  Interventions: Device: Moria M2 microkeratome (MK)
- femtosecond group (Other): 30 eyes were treated by femtosecond laser
  Interventions: Device: Visumax femtosecond laser

INTERVENTIONS:
Device: Visumax femtosecond laser
  Arms: femtosecond group
Device: Moria M2 microkeratome (MK)
  Arms: microkeratome group

SUMMARY:
this is an interventional prospective clinical study which was conducted to evaluate the efficacy, safety, predictability, ocular aberrations, and flap thickness predictability of Visumax femtosecond laser (FSL) compared to Moria M2 microkeratome (MK) in mild to moderate myopia.

DETAILED DESCRIPTION:
This study included 60 eyes who were divided into two groups. Thirty eyes in group (I) in which the flap was created with Visumax FSL, while in group II (30 eyes) the Moria M2 MK was used. Keratometric, refractive, and aberrometric measurements were compared preoperatively and 3 months postoperatively. The intraoperative subtraction pachymetry (the SP 100 Handy pachymeter (Tomey, Nagoya, Japan) was used for preoperative pachymetry and flap thickness measurement.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients were eligible for the study if they were older than 18 years and younger than 40 years.
* Stable myopia up to -6.0D and astigmatism up to -3.0D determined by manifest refraction for at least 6 months.
* best corrected distance visual acuity of at least 20/20, and stable keratometry after cessa¬tion of soft contact lens wear for at least 2 weeks.

Exclusion Criteria:

* any anterior seg¬ment pathology.
* any form of retinal degeneration. unstable myopia.
* severe dry eye.
* corneal thickness that would have resulted in less than 300 µm residual stromal thickness.
* Patients who had keratoconus or were keratoconus suspects.
* previous ocular sur¬gery.
* a history of herpes zoster ophthalmicus or herpes simplex keratitis.
* a history of a steroid-responsive rise in in¬traocular pressure (IOP) or a preoperative IOP of more than 21 mmHg.
* diabetes mellitus, autoimmune dis¬ease, connective tissue disease, and chronic use of systemic corticosteroid or immunosuppressive therapy were also excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-05-29 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
visual outcomes | 6 months
  uncorrected and best corrected distant visual acuity in LogMAR
refractive outcomes | 6 months
  sphere in diopter, cylinder in diopter cylinder and spherical equivalent in diopter

CONTACTS AND LOCATIONS:
Overall Officials: Magda Torky, Principal Investigator — daralshifa hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torky MA, Al Zafiri YA, Khattab AM, Farag RK, Awad EA. Visumax femtolasik versus Moria M2 microkeratome in mild to moderate myopia: efficacy, safety, predictability, aberrometric changes and flap thickness predictability. BMC Ophthalmol. 2017 Jul 17;17(1):125. doi: 10.1186/s12886-017-0520-5. PMID 28716114